CLINICAL TRIAL: NCT01639755
Title: European New Texture Implant Clinical Experience With Shaped Breast Implants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ENTICE-002
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Breast Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Al participants who had new texture shaped breast implants surgically implanted.
  Interventions: Device: new texture shaped breast implants

INTERVENTIONS:
Device: new texture shaped breast implants — breast implant surgery

SUMMARY:
The purpose of this study is to obtain clinical experience with the use of new texture, shaped breast implants in bilateral primary breast augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to undergo bilateral breast augmentation with subglandular, submuscular, or biplanar placement of the breast implants by inframammary approach only
* Be a candidate for the device styles and sizes available in the study

Exclusion Criteria:

* Have tuberous breasts, congenital anomalies of the breast (e.g., Poland's Syndrome), or grade 3 ptosis
* Have undergone any previous breast surgery
* Have tissue covering determined inadequate or unsuitable by the surgeon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2013-01-30 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Heden, Study Director — Allergan
Locations (2):
- Sweden (2):
  - Klinik 34, Göteburg
  - Akademikliniken 10, Stockholm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 19
Completed | 0
Not Completed | 19
Not completed — Study Ongoing | 15
Not completed — Patient had device explantation | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator Overall Satisfaction With the Device Using a 5-Point Scale
Description: The investigator evaluated the overall satisfaction with the device using a 5-point scale where 1=definitely dissatisfied with the device to 5=definitely satisfied with the device.
Time Frame: 3 months
Population: Full analysis population included all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 19
score on a scale | 4.6 (0.77)

2. Secondary Outcome: Subject Satisfaction With Breasts Using the BREAST-Q Questionnaire
Description: Participants evaluated satisfaction with their breasts using the BREAST-Q. Summary scores were computed by summing the score of each response and transferring them to a 0 (worst) to 100 (best) scale.
Time Frame: 6 months
Population: Full analysis population included all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 19
score on a scale | 87.1 (16.95)

3. Secondary Outcome: Investigator Evaluation of Whether the Implant is Palpably Distinguishable From the Tissue
Description: The investigator examined the breasts and evaluated whether the implant was palpably distinguishable from the tissue using a 5-point scale where 1=implant very easy to distinguish from the tissue to 5=implant indistinguishable from the tissue.
Time Frame: 6 months
Population: Full analysis population included all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 19
score on a scale | 2.5 (0.77)

4. Secondary Outcome: Percentage of Participants With Capsular Contracture Evaluated by Four-Grade Baker Scale
Description: The investigator evaluated capsular contracture (lining of cells formed around the device as the body's response to a foreign object) using the Four-Grade Baker scale where: Grade I= Breast is normally soft and looks natural, Grade II= Breast is a little firm but looks normal, Grade III=Breast is firm and looks abnormal or Grade IV= Breast is hard, painful, and looks abnormal. The percentage of participants in each Baker Grade is reported.
Time Frame: Interim analysis: 12 months
Population: Participants from the Full Analysis population with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 18
percentage of participants
  Baker Grade I | 88.9
  Baker Grade II | 11.1
  Baker Grade III | 0.0
  Baker Grade IV | 0.0

5. Secondary Outcome: Percentage of Participants With Local Complications
Description: The percentage of participants experiencing local complications (in the area of the implant) is reported.
Time Frame: Interim analysis: 12 months
Population: Full analysis population included all participants.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 19
percentage of participants
  Breast pain | 100.0
  Implant malposition | 15.8

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=19)
Device dislocation (General disorders) | 2
Anxiety (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=19)
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Breast complication associated with device (General disorders) | 1
Helicobacter gastritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 19
Nervous system disorder (Nervous system disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.